CLINICAL TRIAL: NCT00105248
Title: Multidimensional Intervention Program to Reduce Antibiotic Prescriptions for Acute Respiratory Tract Infections in Adults: a Randomized Controlled Trial in Primary Care
Brief Title: Patient Centered Communication Training to Reduce Antibiotic Use in Acute Respiratory Tract Infections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Basel Institute of Clinical Epidemiology (BICE) (Other); Swiss National Science Foundation (Other); Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 3200B0-102137; 04B29; 2003/051; 242/03
Record Dates: First submitted 2005-03-10; First posted 2005-03-11 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-05

CONDITIONS: Respiratory Tract Infections
Keywords: acute repiratory infections; antibiotic therapy; patient-centred communication; randomized controlled trial
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: patient-centered communication training

SUMMARY:
The purpose of this study is to evaluate the effectiveness of a short training program for general practitioners in patient-centered communication to reduce antibiotic prescription for acute respiratory tract infections (ARTI).

DETAILED DESCRIPTION:
Acute respiratory tract infections (ARTI) constitute the most frequent reason for seeking ambulatory care and for the prescription of antibiotics, despite the mostly viral origin of ARTI. Antibiotic prescriptions for ARTI increase unnecessary drug expenditures and are the main reason for increasing drug resistance of common bacteria. Evidence from intervention studies shows that merely providing physicians with guidelines and educational material for the management of acute respiratory tract infections is not enough to reduce antibiotic prescriptions for these conditions. The main reasons for antibiotic prescription in ARTI are non-medical and related to the physician patient relationship, patients' expectations and beliefs about the benefit of antibiotics. Therefore patient-centered communication could be a promising approach to reduce the rate of antibiotic prescription in ambulatory care.

Comparison: General practitioners (GPs) trained in patient-centered communication in addition to evidence-based guidelines for diagnosis and treatment of ARTI compared to GPs just introduced to evidence-based guidelines.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Symptoms of an acute respiratory tract infection for >1 and <28 days

Exclusion Criteria:

* Patients without informed consent
* Not fluent in German
* Patients with a psychiatric disorder
* Patients with a recurrent respiratory system infection with antibiotic treatment in the previous 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900
Dates: Start 2004-01; Study Completion 2004-06

PRIMARY OUTCOMES:
Up-take of antibiotic prescription confirmed by pharmacists within 2 weeks following the initial consultation

SECONDARY OUTCOMES:
Patient satisfaction with consultation (on validated scale)
patient enablement (on validated scale)
days with restriction from ARTI within 14 days initial consultation
side effects from medication
re-consultation rates
days off from work

CONTACTS AND LOCATIONS:
Overall Officials: Heiner Bucher, Prof., Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- Basel institute for clinical epidemiology, Basel, Switzerland